CLINICAL TRIAL: NCT02772224
Title: The Efficacy and Safety of Paclitaxel-eluting Balloons for the Treatment of Below the Knee Peripheral Arterial Disease as Compared to Conventional Balloon Angioplasty: a Randomized Controlled Clinical Trial.
Brief Title: Efficacy and Safety of Paclitaxel-eluting Balloons for Below the Knee Peripheral Arterial Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Maoquan Li, Prof. Dr.Li, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 425008534
Record Dates: First submitted 2016-05-08; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug eluting balloon angioplasty (Experimental): Paclitaxel coated balloon angioplasty
  Interventions: Device: Drug eluting balloon angioplasty
- Conventional balloon angioplasty (Active Comparator): Conventional balloon angioplasty
  Interventions: Device: Conventional balloon angioplasty

INTERVENTIONS:
Device: Drug eluting balloon angioplasty — In the DEB group, the guide wire will be passed through the occluded or stenosed lumen and the predilatation of the target lesion with standard balloon(s) will be performed before dilatation with a paclitaxel-eluting balloon of the diameter, at least about that of the pre-dilatation balloon (Arteryguard, Rientech, Dezhou, China). The drug eluting balloons will then be inflated according to the manufacturer recommendations. The patients will then be followed every six months for a year to compare its treatment efficacy and safety with that of conventional balloon angioplasty group.
  Arms: Drug eluting balloon angioplasty
Device: Conventional balloon angioplasty — The guide wire will be passed through the occluded or stenosed lumen and the conventional balloons will be inflated as recommended by the manufacturer. The primary and secondary outcome will then be assessed and compared with DEB group, on follow up at six and 12 months.
  Arms: Conventional balloon angioplasty

SUMMARY:
Comparing the efficacy and safety of drug-eluting balloons (DEB) for the treatment of below-the-knee peripheral arterial occlusive disease with conventional balloon angioplasty (BA).

DETAILED DESCRIPTION:
Over the past decade, percutaneous transluminal angioplasty (PTA) has established its position in the treatment of below the knee arterial occlusive disease with intermittent claudication and/or critical limb ischemia. However, the efficacy of percutaneous transluminal angioplasty (PTA) with conventional balloons, is limited by the high 12-month restenosis and target lesion revascularization (TLR) rates. Local delivery of newer anti-proliferative drug via drug-eluting balloons (DEBs) has recently shown promising results in the treatment of femoropopliteal disease, and in the BTK area, a reduction in 3-month binary restenosis has been observed compared with historical controls treated with PTA. Drug eluting balloon has three potential advantages: (1) homogenous drug transfer to the vessel wall; (2) highest drug concentrations at the vessel wall at the time of injury; and (3) absence of a stent or delivery polymer.

This study sought to investigate the long-term efficacy and safety of new drug (Paclitaxel)-eluting balloons (DEB) for the treatment of below the knee peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Peripheral vascular disease with or without diabetes.
2. Rutherford class 2-6.
3. Target lesions with a diameter reduction of at least 50% on angiography, and without past history of any intervention.
4. Target vessel with 2.0--10.0mm in diameter and having a lesion of about 4cm-20cm in length.
5. Written informed consent signed by the patients or representatives

Exclusion Criteria:

1. Previous bypass surgery or stent placement at the ipsilateral lower limb
2. History of intolerance to antiplatelet therapy, heparin, or contrast media.
3. Bleeding diathesis;
4. Active systemic bacterial infection;
5. Severely impaired renal function (serum creatinine level > 2.5 mg/dL.
6. Expected survival time of less than 24 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate | 12 months
  The primary study endpoint was the occurrence of > 50% of restenosis in the treated vessel after 12 months as assessed by digital substraction angiography (DSA).
Peak systolic velocity ratio | 12 months
  Peak systolic velocity ratio ≥ 2.4 by Doppler's ultrasonography was the end point of the study for the patient who did not undergo angiography after 12 months.

SECONDARY OUTCOMES:
Rutherford scale | Immediately after procedure
  Clinical success is to be defined as an improvement in Rutherford scale of at least one category after the procedure.
ABI value | Immediately after procedure
  Hemodynamic success is to be defined as an improvement of ABI value by ≥ 0.1 after the procedure and lack of deterioration > 0.15 in relation to the maximal value recorded before the procedure.
Residual stenosis | Immediately after procedure
  The technical success of the procedure is to be defined as PTA of a lesion with >30 % residual stenosis and lack of flow rate-limiting dissection immediately after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth people's hospital, Tongji university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liistro F, Porto I, Angioli P, Grotti S, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for below the knee angioplasty evaluation (DEBATE-BTK): a randomized trial in diabetic patients with critical limb ischemia. Circulation. 2013 Aug 6;128(6):615-21. doi: 10.1161/CIRCULATIONAHA.113.001811. PMID 23797811
- [Result] Karnabatidis D, Spiliopoulos S, Katsanos K, Siablis D. Below-the-knee drug-eluting stents and drug-coated balloons. Expert Rev Med Devices. 2012 Jan;9(1):85-94. doi: 10.1586/erd.11.67. PMID 22145843
- [Result] Jens S, Conijn AP, Koelemay MJ, Bipat S, Reekers JA. Randomized trials for endovascular treatment of infrainguinal arterial disease: systematic review and meta-analysis (Part 2: Below the knee). Eur J Vasc Endovasc Surg. 2014 May;47(5):536-44. doi: 10.1016/j.ejvs.2014.02.012. Epub 2014 Mar 17. PMID 24650395
- [Result] Schnorr B, Albrecht T. Drug-coated balloons and their place in treating peripheral arterial disease. Expert Rev Med Devices. 2013 Jan;10(1):105-14. doi: 10.1586/erd.12.67. PMID 23278227
- [Result] Zeller T, Baumgartner I, Scheinert D, Brodmann M, Bosiers M, Micari A, Peeters P, Vermassen F, Landini M; IN.PACT DEEP Trial Investigators. IN.PACT Amphirion paclitaxel eluting balloon versus standard percutaneous transluminal angioplasty for infrapopliteal revascularization of critical limb ischemia: rationale and protocol for an ongoing randomized controlled trial. Trials. 2014 Feb 19;15:63. doi: 10.1186/1745-6215-15-63. PMID 24552184